CLINICAL TRIAL: NCT05668845
Title: Paragastric Autonomic Neural Blockade as Part of Combined Anesthesia. Impact on Anesthetic Agents Consumption: A Randomized Clinical Trial Protocol
Brief Title: Paragastric Autonomic Neural Blockade as Part of Combined Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Simón Bolívar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-CEI-USB-CE-0394-01; PRO-CEI-USB-CE-0394-02 (Other: Unisimon)
Record Dates: First submitted 2022-11-26; First posted 2022-12-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Opioid Use; Anesthesia Morbidity
Keywords: Autonomic; Blockade; Opioids; Anesthetics; Recovery time

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: The patient and the independent investigator assessing and recording the patient's data will be blinded to treatment arm assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PG-ANB performed at the outset of LSG (Experimental): PG-ANB is performed early in the procedure as a first step before starting the sleeve gastrectomy.
  Interventions: Other: PG-ANB performed at the outset of LSG
- PG-ANB performed at the end of LSG (Active Comparator): PG-ANB is performed at the end of the sleeve gastrectomy
  Interventions: Other: PG-ANB performed at the end of the LSG

INTERVENTIONS:
Other: PG-ANB performed at the outset of LSG — The paragastric lesser omentum neural block is performed with a 25-gauge needle attached to a venous catheter extension introduced through the left 12-mm port. The needle is capped during its introduction, and the cap is removed inside the abdomen using a grasper and kept under direct vision. Infiltration of 20 mL of non-diluted 0.5% bupivacaine is performed at six levels with careful aspiration preceding fluid infiltration. Four areas are adjacent to the vagus nerves and branches, and two are in the vicinity of the common hepatic and left gastric arteries. This is performed at the outset of the LSG.
  Arms: PG-ANB performed at the outset of LSG
Other: PG-ANB performed at the end of the LSG — The paragastric lesser omentum neural block is performed with a 25-gauge needle attached to a venous catheter extension introduced through the left 12-mm port. The needle is capped during its introduction, and the cap is removed inside the abdomen using a grasper and kept under direct vision. Infiltration of 20 mL of non-diluted 0.5% bupivacaine is performed at six levels with careful aspiration preceding fluid infiltration. Four areas are adjacent to the vagus nerves and branches, and two are in the vicinity of the common hepatic and left gastric arteries. This is performed at the end of the LSG>
  Arms: PG-ANB performed at the end of LSG

SUMMARY:
To evaluate the effect of early autonomic blockade on the consumption of remifentanil and halogenated anesthesia in the intraoperative period during laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Balanced general anesthesia, even if combined with local anesthesia or parietal blocks such as transversus abdominis plane (TAP), subcostal, or pararectal blocks, is insufficient to block the autonomic impulses released during most intra-abdominal visceral surgeries, especially in laparoscopic sleeve gastrectomy (LSG). These impulses are, in part, responsible for the hemodynamic changes observed during different phases of LSG and the subsequent visceral pain and associated symptoms, such as nausea and vomiting, observed in a substantial number of patients in the immediate postoperative period after LSG and other minimally invasive procedures. Visceral pain substantially impacts patients' quality of life, recovery time, nursing time allocation, and resultant risk of opioid abuse. Nausea, food intolerance, and pain are responsible for most readmissions after LSG and other bariatric procedures. Many of these patients have associated severe respiratory impairments and other comorbidities. They often need increased amounts of halogenated anesthetics, opioid analgesics, antiemetics, and other anesthetic modalities such as epidural anesthesia. A recent randomized clinical trial (RCT) demonstrated that a novel approach, namely paragastric autonomic neural blockade (PG-ANB), is safe and effective in addressing visceral pain while reducing the need for analgesics, including opioids and the decreasing nausea and vomiting in the first 24 hours after a laparoscopic sleeve gastrectomy. In an observational series, we found that by performing PG-ANB as the first step in LSG, the need for morphine-equivalent doses and halogenated anesthetics diminished, and hemodynamic stability increased while maintaining the previously reported reduction of postoperative visceral pain and associated symptoms. Similarly, when implementing a variation of the autonomic blockade targeting proper pathways as an early step in cholecystectomy, the same beneficial effects were observed in affected patients.

ELIGIBILITY:
Inclusion Criteria:

-all adult patients scheduled for LSG at each participating institution.

Exclusion Criteria

* the inability to perform a PG-ANB because of anatomical difficulties
* the need for revisional surgery
* the need for concomitant hiatal hernia repair or other surgical procedures
* conversion to open surgical procedures
* allergies to local anesthetics or medication described in the anesthesia protocol
* intraoperative complications (e.g., visceral or vascular perforations)
* anesthesia-related complications requiring admission to intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative Remifentanil consumption | duration of the anesthesia
  The amount of remifentanil administered will be calculated based on the amount of the consumed mix and reported as total mcg and mcg/kg/min.
Intraoperative consumption of the halogenated agent (sevoflurane) | duration of the anesthesia
  The anesthetic machine will determine the administered amount of sevoflurane (Dräger Primus) which will be reported in ml/min.

SECONDARY OUTCOMES:
recovery from anesthesia measured by the Modified Aldrete Scale | one hour after surgery
  The Modified Aldrete scale from 0 to 15 (a higher score correlates with better recovery from anesthesia) will be assessed and recorded 15 minutes and 1 hour after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pantoja, MD, Study Chair — Universidad Simón Bolívar
Locations (1):
- clinicas Portoazul e Iberoamerica, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617
- [Derived] Daes J, Pantoja R, Luquetta J, Luque E, Hanssen A, Rocha J, Morrell DJ. Impact on Anesthetic Agent Consumption After Autonomic Neural Blockade as Part of a Combined Anesthesia Protocol: A Randomized Clinical Trial. Anesth Analg. 2024 Sep 1;139(3):581-589. doi: 10.1213/ANE.0000000000006769. Epub 2023 Dec 13. PMID 38091501